CLINICAL TRIAL: NCT06551233
Title: A Clinical Study on the Safety and Efficacy of 9MW2821 in Patients With High-risk Non-muscle-invasive Bladder Cancer (NMIBC) That Have Previously Failed to Intravesical Therapy
Brief Title: Safety and Efficacy of 9MW2821 in the Treatment of High-risk Non-muscle-invasive Bladder Cancer (NMIBC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-UC-107
Record Dates: First submitted 2024-04-23; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation and expansion (Experimental): Induction period: once a week, 6 times in total. Maintenance period: once per 28 days, 9 times in total. Intravesical therapy
  Interventions: Drug: 9MW2821

INTERVENTIONS:
Drug: 9MW2821 — Patients will be evaluated from low dose to high dose through intravesical therapy and then select the suitable doses to expand according to study data.

SUMMARY:
Assess the safety and efficacy of 9MW2821 in patients with high-risk non-muscle-invasive bladder cancer (NMIBC) who have previously failed to intravesical therapy. Provide a new treatment option for patients with NMIBC recurrence, reduce the risk of tumor recurrence, decrease the rate of radical bladder surgery, and enhance the quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old before signing the informed consent.
* Subjects must have previously failed to at least one kind of intravesical therapy, including but not limited to BCG, gemcitabine, etc.
* Subjects refuse or are intolerant to BCG therapy.
* Subjects must have completed a standard TURBT surgery within 6 weeks before the first dose of the study drug and have no evidence of residual tumors in the surgical field.
* Tumor tissue samples from TURBT must be provided (≥5 slides), along with relevant pathological reports.
* Histological and pathological diagnosis of urothelial carcinoma (with a major component >50%) , with the confirmation of no-muscle invasion.
* Subjects must be categorized as high-risk NMIBC
* Subjects refuse or are intolerant to radical cystectomy.
* Clinical non-metastatic bladder cancer (N0, M0) determined by CT scan.
* Adequate function of heart, bone marrow, liver, and kidney.
* ECOG 0-1
* Subjects must be willing to take highly effective contraception during the study and 180 days after the last dose of 9MW2821 (a negative serum pregnancy test result within ≤7 days before enrollment for the female).

Exclusion Criteria:

* History of muscle invasive or metastatic bladder cancer.
* History of other malignancies within 3 years.
* Other systemic anti-cancer therapies within 3 weeks before the first dose of the study drug.
* Surgery (such as TURBT) or radiotherapy for bladder lesions within 2 weeks before the first dose.
* Hypersensitivity reactions to certain components of 9MW2821 or similar drugs.
* Persistence of adverse reactions caused by prior anti-tumor therapy before the first dose, does not recover to grade 1 and below, according to NCI-CTCAE v5.0.
* Active systemic infections that require treatments within 7 days before the first dose.
* Severe cardiovascular diseases within 6 months before the first dose.
* History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
* History of autoimmune diseases.
* Serum virology tests: positive results for HBsAg or HBcAb, with positive HBV-DNA copies (≥500IU/mL); positive HCV-Ab results, with positive HCV-RNA results; positive HIV-Ab results.
* Prior treatment with drugs targeted Nectin-4 or MMAE-conjugated ADC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | up to 12 months
  assess the incidence of AE/SAE
RP2D and MTD | up to 12 months
  Determine the recommended phase 2 dose (RP2D) and the maximum tolerated dose (MTD) that may occur.

SECONDARY OUTCOMES:
DFS rate of 12 months | Up to 12 months
  Disease-free survival rate of 12 months
DoR of CR | Up to 20 months
  Duration of complete response
CR rate of 3/6/12 months | Up to 12 months
  Complete response rate of 3/6/12 months
DFS | Up to 20 months
  Disease-free survival
Duration to radical cystectomy | Up to 20 months
  Duration to radical cystectomy
Proportion of radical cystectomy | Up to 20 months
  Proportion of radical cystectomy
Biomarker parameter | Up to 20 months
  Expression of Nectin-4

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China